CLINICAL TRIAL: NCT00937430
Title: Bowel Preparation and Return of Bowel Function After Pelvic Organ Prolapse Surgery.
Brief Title: Bowel Preparation and Pelvic Organ Prolapse Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 09001
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Bowel preparation
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bowel preparation group (Experimental): Patients randomized to this arm will perform a bowel preparation prior to their pelvic organ prolapse surgery.
  Interventions: Other: Bowel preparation (Fleets enema)
- No Bowel preparation group (No Intervention): Patients randomized to this group will not be performing a bowel preparation prior to their pelvic organ prolapse surgery.

INTERVENTIONS:
Other: Bowel preparation (Fleets enema) — Use of Bowel preparation (Fleets enema)
  Arms: Bowel preparation group

SUMMARY:
The purpose of this study is to find out if performing a bowel preparation prior to pelvic organ prolapse surgery has any effect on the return of bowel function after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 21-90 years.
* Have a posterior vaginal wall prolapse.
* Are undergoing vaginal prolapse reconstructive surgery including posterior repair with suspension of the vaginal apex (top) to the ligaments in your pelvis, repair of the cul de sac or "enterocele", with or without anti-incontinence surgery.
* Are receiving general anesthesia.

Exclusion Criteria:

* Patient undergoing concomitant anal sphincteroplasty, rectovaginal fistula repair, rectopexy, or rectal resection/reanastomosis.
* Patient undergoing any mesh augmentation.
* Patient with any neurological condition involving bowel function.
* Patient on regular narcotic medication preoperatively.
* Patient does not want to be in the group she was randomized to.
* Patient currently pregnant or planning to become pregnant, or breastfeeding.
* Patient with ascites.
* Patient with known or suspected gastrointestinal obstruction or perforation.
* Patient with history of hyperparathyroidism.
* Patient with dehydration.
* Patient with active inflammatory bowel disease.
* Patients with congestive heart failure.
* Patients with dialysis dependent renal disease.

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Measure the return of bowel function after pelvic organ prolapse surgery. | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel N Pauls, M.D., Study Director — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States